CLINICAL TRIAL: NCT05898763
Title: T-cell Epitopes Associated With Impaired Peptide Processing (TEIPP)- Targeting Immunotherapy in Patients With Relapsed Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: TEIPP Immunotherapy in Patients With NSCLC
Acronym: TEIPP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Joachim Aerts, MD PhD, Principal Investigator (MD PhD), Erasmus Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL75654.000.20
Record Dates: First submitted 2023-04-24; First posted 2023-06-12 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immunotherapy; Palliative treatment; Dose-escalation study; Checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — montanide ISA 51; pembrolizumab

STUDY DESIGN:
Intervention Model Description: A multicenter, open label non-randomized phase I/II dose escalation study with extension cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients will be vaccinated with the TEIPP24 vaccine in Montanide ISA 51 every three weeks for a total of three rounds of vaccination. The total treatment duration is 9 weeks for each patient. The three dose levels tested are 20, 40 and 100 µg of peptide. Dose 1: 20 µg of peptide in Montanide ISA 51; Dose 2: 40 µg of peptide in Montanide ISA 51; Dose 3: 100 µg of peptide in Montanide ISA 51. Patients in the extension cohort will receive the highest safest dose of peptide in combination with pembrolizumab.
  Interventions: Drug: TEIPP24 (LRPAP7-30V-SLP vaccine in Montanide ISA-51)

INTERVENTIONS:
Drug: TEIPP24 (LRPAP7-30V-SLP vaccine in Montanide ISA-51) — Patients will receive three rounds of vaccination three weeks apart via one subcutaneous (SC) injection in an alternating limb. Patients in the extension cohort will receive the highest safest dose in combination with pembrolizumab (a CPI).These patients will receive three rounds of combination treatment with TEIPP24 vaccination and pembrolizumab every three weeks. Pembrolizumab will be administered as per standard of care.
  Other Names: Pembrolizumab

SUMMARY:
In this multicenter, open label non-randomized phase I/II dose escalation study with extension cohort HLA-A*0201-positive patients with non small cell lung cancer (NSCLC) can be included. The primary aim of this study is determine the safety, tolerability and immune modulating effects of the therapeutic LRPAP1 synthetic long peptide (LRPAP7-30V-SLP) vaccine (TEIPP24) at different doses. Secondary objectives are to assess the specificity and immune modulatory effects of the vaccine, to assess the antigen and immune status of the patients, and to determine progression free survival (PFS), overall survival (OS), and the radiological tumor response up to one year after first vaccination.

DETAILED DESCRIPTION:
Immunogenic tumors can be controlled by tumor-reactive Tcells either directly or after checkpoint blockade. In the end, most tumors will develop mechanisms to escape immune control. One of such a mechanism is formed by the functional impairment of the intracellular peptide transporter TAP1/TAP2 by mutation of downregulated expression. As a result the presentation of conventional T-cell epitopes in HLA class I is lost, and hence tumor-reactive CD8+ T-cells fail to recognize and kill tumor cells. This type of immune escape can occur in up to 50% of primary tumors and is increased in the metastatic lesions of such tumors. The presence of these TAP defects correlate with worse clinicopathological parameters and has been associated with loss of durable benefit to checkpoint inhibition. The unmet need, therefore, is the development of a therapy that can reinforce effective tumor-immunity to cancers displaying TAP-defects for which conventional therapeutic cancer vaccines and/or checkpoint blockade do not work. TEIPP therapy may fill this position by reinstalling an effective antitumor response to TAP-defective tumors thereby increasing the overall survival of patients failing first line therapy.

In this prospective, single arm, multicenter, open-label, phase I-II clinical study, HLA-A*0201-positive patients with NSCLC failing first line of treatment will be enrolled in 3 cohorts and one extension cohort of 6 patients (at the highest safe and tolerable dose) combined with a checkpoint inhibitor targeting PD-1/PD-L1 (CPI), to include 24 patients in total. The maximal total treatment duration is 9 weeks. The first 6 patients will be enrolled in cohort 1, the next 6 patients in cohort 2, the next 6 patients in cohort 3. The decision to start enrollment at the next dose level will be made by assessing the safety after 3 out of 6 patients at the previous dose level have completed vaccine therapy.

Patients will receive an off the shelf TEIPP24 vaccine mixed with Montanide ISA-51 adjuvant, which will be administered every three weeks for a period of three rounds of vaccination. Patient cohort 1 will be treated with TEIPP24 at a dose of 20ug of peptide, patients in cohort 2 with TEIPP24 at a dose of 40ug of peptide and patients in cohort 3 with TEIPP24 at a dose of 100ug of peptide. Patients in the extension cohort will receive the highest safest dose in combination with pembrolizumab (a CPI). Patients will receive three rounds of vaccination three weeks apart via one subcutaneous (SC) injection in a limb. The SC route of administration of TEIPP24 vaccine is dictated by the use of Montanide ISA51. Subsequently patients will be followed up to 1 year after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Pathologically and radiologically confirmed advanced NSCLC.
* Progression after minimally 4 cycles of combination platinum containing chemotherapy and immunotherapy (PD1), or after 4 cycles of platinum containing chemotherapy and immunotherapy (PD-1) followed by maintenance chemo immunotherapy
* HLA-A*0201 positive
* An expected survival of at least 3 months
* WHO/ECOG performance status ≤ 2 (Appendix 3)
* Adequate renal function as defined by creatinine clearance > 40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR)
* Adequate hepatic function as evidenced by

  * Serum total bilirubin ≤ 2.5 × upper limit of normal (ULN) unless considered due to hepatic metastases
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to hepatic metastases
* Ability to return to the hospital for adequate follow-up as required by this protocol.
* Written informed consent according to International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) .

Exclusion Criteria:

* Active infection, including hepatitis B or C or HIV infection that is uncontrolled at inclusion. An infection controlled with an approved or closely monitored antibiotic/antiviral/antifungal treatment is allowed.
* Current use of steroids (or other immunosuppressive agents). Patients must have had 6 weeks of discontinuation and must stop any such treatment during the time of the study. Prophylactic usage of dexamethasone during chemotherapy is excluded from this 6 weeks interval.
* Concomitant participation in another clinical intervention trial (except participation in a biobank study).
* Pregnant or lactating women.
* Known allergy to any of the ingredients of the vaccine (peptide, Montanide ISA-51, trifluoroacetic acid, acetonitrile, dichloromethane, dimethylsulfoxide).
* Any medical or psychological condition deemed by the Investigator to be likely to interfere with a patient's ability to give informed consent or participate in the study
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Patients with a currently active second malignancy. However, patients with the following history/concurrent conditions are allowed: Basal or squamous cell carcinoma of the skin; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histologic finding of prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Safety assessment based on the incidence rate of serious adverse drug reactions (ADR) as assessed by NCI-CTCAE version 5.0. | Week 8 (two weeks after the third TEIPP24 vaccination)
  Safety of the therapeutic LRPAP1 synthetic long peptide ( LRPAP7-30V-SLP) vaccine (TEIPP24) determined by the incidence rate at each dose level based on the following safety parameters: adverse drug reactions (ADR) and serious ADRs, changes in haematology and chemistry values, including those associated with hepatic and renal function, and assessment of physical examinations, vital signs and performance status. NCI-CTCAE version 5.0 will be used.
Tolerability assessment based on patients' tolerability of adverse drug reactions (ADR) | Week 8 (two weeks after the third TEIPP24 vaccination)
  Tolerability of the therapeutic LRPAP1 synthetic long peptide ( LRPAP7-30V-SLP) vaccine (TEIPP24) determined by patients' tolerability of ADRs. NCI-CTCAE version 5.0 will be used.
Immunogenicity assessed by HLA-A*0201-restricted LRPAP21-30 -specific CD8+ T-cell reactivity | Week 3-6-9 (three weeks after every TEIPP24 vaccination)
  HLA-A*0201-restricted LRPAP21-30 -specific CD8+ T-cell reactivity will be determined by measuring the magnitude and function of HLA-A*0201-restricted LRPAP21-30 -specific CD8+ Tcells present in the blood and/or tumor samples before and after TEIPP24 vaccination at different dose levels.

SECONDARY OUTCOMES:
The specificity and immune modulatory effect of the vaccine, determined by isolating LRPAP(21-30V)-specific CD8+ T cells | Week 3-6-9 (three weeks after every TEIPP24 vaccination)
  The specificity and immune modulatory effect of the vaccine is determined by isolating LRPAP(21-30V)-specific CD8+ T cells that are cocultured with tumor cells. CD8+ T cells that recognize LRPAP presented on these tumor cells will produce type 1 cytokines which is measured by ELISA.
Immunohistochemical staining of tumor material | Before (week 0) and after treatment (week 9)
  The pretreatment (and when available post-vaccination) tumor material will be subjected to immunohistochemical staining for TAP 1, TAP 2, HLA class I and LRPAP.
Progression free survival (PFS) | From week 0 up to week 52
  Progression free survival (PFS) defined as the time frame between the first vaccination and date of progression
Overall survival (OS) | From week 0 up to week 52
  Overall survival (OS) defined as the time frame between the first vaccination and date of death
Radiological tumor response | From week 0 up to week 52
  To determine the radiological tumor response up to one year after first vaccination according to RECIST v.1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No